CLINICAL TRIAL: NCT04382222
Title: Sensitivity and Accuracy of Prenatal Diagnosis of Severe Congenital Heart Diseases in the Antwerp Region
Brief Title: Prenatal Screening for Congenital Heart Diseases in the Antwerp Region
Acronym: SEC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Prof Yves Jacquemyn, Professor, Universiteit Antwerpen
Other Study IDs: 20/16/205 - 001126
Record Dates: First submitted 2020-05-06; First posted 2020-05-11 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Congenital Heart Disease in Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: prenatal ultrasound — prenatal cardiac ultrasound

SUMMARY:
No systematic research has been done in the last 15 years on the accuracy of prenatal ultrasound of congenital heart diseases in Belgium. Nor are there any population-based studies available on this subject for Belgium. Based on the data of EUROCAT (European Surveillance of Congenital Anomalies) the investigators analyse prenatal diagnostic sensitivity of congenital heart diseases in the EUROCAT regions Antwerp (Flanders, Belgium)

DETAILED DESCRIPTION:
Congenital heart defects are a leading cause of infant mortality with an incidence of 0,4-1,3% at birth. Although prenatal detection rates vary widely, morphological (structural) cardiac malformations are among the most frequently missed abnormalities by prenatal ultrasonography.

However, identifying fetal cardiac abnormalities early in pregnancy is essential. Early diagnosis allows extensive cardiac ultrasound, genetic testing and planning delivery in a paediatric-cardiac centre offering optimal neonatal care.

It also may allow the future parents to consider and decide for a termination of pregnancy in case of a severe fetal heart malformation with poor prognosis.

The investigator conducts a retrospective study on 2500 cases of congenital heart diseases over 20 years. Detailed data for this were made available by the EUROCAT Antwerp registry, a population-based database with controlled, reliable and robust data.

The study wants to reveal the prevalence and prenatal diagnostic sensitivity of congenital heart defects in the EUROCAT regions Antwerp (Flanders) and especially the evolution of the prenatal diagnostic rate over time.

In the second phase, a similar study in two adjacent regions, Hainaut (Wallonia, Belgium) and Groningen (The Netherlands) will follow.

On condition of correct statistic processing, these data will be suitable to compare the prevalence and to benchmark diagnostic rates of congenital heart defects in these three regions.

ELIGIBILITY:
Inclusion criteria

* All fetal congenital heart diseases registered in the Antwerp-EUROCAT database,
* In the period 1/1/1997-31/12/2017 period

Exclusion criteria

* All cases of congenital heart diseases where the mother was under <18 years old.
* All cases of congenital heart diseases were the parents did not allow inclusion in the EUROCAT registered.
* All cases of congenital heart diseases where the mother delivered outside the EC countries.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Low risk pregnancies
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
sensitivity and accuracy of prenatal ultrasound for cardiac malformations | retrospective 20 years
  retrospective analysis of prenatally missed and diagnosed congenital heart disaeses iseaersa

CONTACTS AND LOCATIONS:
Overall Officials: Paul Ramaekers, MD, Study Chair — University Antwerpen; Yves Jacquemyn, Study Chair — University Antwerpen
Locations (1):
- University Hospital Antwerp, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No